CLINICAL TRIAL: NCT01328210
Title: Effects of Blood Letting on Insulin Sensitivity and Blood Pressure in Patients With Metabolic Syndrome: A Randomized Controlled Trial
Brief Title: Effects of Blood Letting in Metabolic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other); University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Professor of Medicine, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2006-AV
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; Phlebotomy; blood letting; hypertension; insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Insulin Resistance | interventions — Bloodletting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- blood letting (Experimental): Blood letting was performed immediately after baseline assessment and after 4 weeks. First blood removal consisted of 400ml, second blood removal was tailored according to subsequent serum ferritin levels between 300- 400 ml.
  Interventions: Procedure: blood letting
- waiting list control (No Intervention): This group received no specific treatment but was offered treatment after termination of the 6-week study phase

INTERVENTIONS:
Procedure: blood letting — blood letting twice within 4 weeks. First blood removal baseline with 400ml of venous blood and second blood removal with 300-400ml according to serum ferritin levels.
  Arms: blood letting

SUMMARY:
Metabolic syndrome (MS) has an increasing prevalence worldwide and there is an urgent need for improvement of medical treatment. In traditional medicine phlebotomy (blood letting) is a recommended treatment for subjects with obesity and vascular disease. Recent studies showed that blood letting with iron depletion may improve insulin sensitivity in patients with diabetes mellitus. The investigators aimed to test if traditional blood letting has beneficial effects in patients with MS. A randomized trial with a sample size of 64 self-referred MS patients was conducted. Patients in the blood letting group were allocated to blood letting intervention and the control group was offered a later treatment (waiting list). In the intervention group 300-400 ml of venous blood were withdrawn at day 1 and after 4 weeks. Primary outcomes were the change of systolic blood pressure and of insulin sensitivity as measured by HOMA-Index.

ELIGIBILITY:
Inclusion Criteria:

* 25-70 years of age
* given diagnosis of metabolic syndrome

Exclusion Criteria:

* clinically significant hepatic, neurological, endocrinologic, or other major systemic or inflammatory disease, including malignancy
* known history of hemochromatosis, or presence of the Cys282Tyr mutation
* history of drug or alcohol abuse
* manifest cardiac disease
* history of disturbances in iron balance (e.g., hemosiderosis from any cause, atransferrinemia)
* preexisting anemia

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | change from baseline at 6 weeks
  Glucose and insulin are measured on the basis of overnight fasting blood samples and Insulin sensitivity calculated according to HOMA-Index
systolic blood pressure | change from baseline at 6 weeks
  Blood pressure is measured twice after 5 minutes rest in the sitting position by sphygmomanometry

SECONDARY OUTCOMES:
diastolic blood pressure | change from baseline at 6 weeks
HbA1c | change from baseline at 6 weeks
blood lipids | change from baseline at 6 weeks
serum ferritin | change from baseline at 6 weeks
adiponectin | change from baseline at 6 weeks
blood count | change from baseline at 6 weeks
serum iron | change from baseline at 6 weeks
hs-CRP | change from baseline at 6 weeks
pulse rate | change from baseline at 6 weeks
serum glucose | change from baseline at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof., M.D., Principal Investigator — Charite-University Medical Centre
Locations (1):
- Kliniken Essen-Mitte, University Duisburg-Essen, Essen, North-Rhine Westfalia, Germany

REFERENCES:
- [Derived] Houschyar KS, Ludtke R, Dobos GJ, Kalus U, Broecker-Preuss M, Rampp T, Brinkhaus B, Michalsen A. Effects of phlebotomy-induced reduction of body iron stores on metabolic syndrome: results from a randomized clinical trial. BMC Med. 2012 May 30;10:54. doi: 10.1186/1741-7015-10-54. PMID 22647517